CLINICAL TRIAL: NCT05645120
Title: Impact of Nutrition Education on Knowledge and Beliefs About Dietary Supplements/Herbal Foods: A Pre - Post Intervention Study
Brief Title: Impact of Nutrition Education on Knowledge and Beliefs About Dietary Supplements/Herbal Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Zeynep Goktas, Principal Investigator, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: GO 21/129
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-12

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: nutrition education; dietary supplements; herbal supplements
MeSH Terms: conditions — Behavior | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Professionals (Experimental): Education intervention for health professionals
  Interventions: Other: Education
- Non-health Professionals (Experimental): Education intervention for non-health professionals
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — All participants attended to a two-part nutrition education program. The education intervention program was administered in two sessions, one week apart. Before the intervention, a pre-test was administered to determine the knowledge and beliefs attitudes of participants. After the pre-test each session consisted of a PowerPoint presentation of about 20 minutes. Education topics included components of adequate-balanced nutrition and its relationship with COVID-19, introduction of food groups, the association between COVID-19 and dietary supplements, herbal foods in the prevention/treatment of COVID-19, considerations regarding DS/HF, food-drug interactions, and COVID-19 drugs and food interactions. The presentation was concluded with the nutritional recommendations for COVID-19. The post-tests were shared with the participants at the end of the second session of the education intervention.

SUMMARY:
A two session nutrition education intervention was administered to health professionals and non-health professionals in separate sessions. Nutrition knowledge status was evaluated with comparing the pre-test and post-test values.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of nutrition education intervention of health professionals and non-health professionals about the effectiveness of dietary supplements/herbal foods (DS/HF) in COVID-19. Study design is a cross-sectional study with an education intervention. This study was conducted through online video communication application. Overall, 106 health professionals and 110 non-health professionals completed the study. The education intervention was administered in two sessions, one week apart for both health professionals and non-health professionals separately. Knowledge level of nutrition and COVID-19 and beliefs about DS/HF in the prevention/treatment of COVID-19 were evaluated with a pre-test and post-test setting. Comparison of the groups before and after the intervention was implemented with the McNemar's test.

ELIGIBILITY:
Inclusion Criteria:

* being 18 to 65 years old
* using social media
* being able to understand Turkish

Exclusion Criteria:

* regular supplement use prior to COVID-19 pandemic
* having a chronic disease that requires dietary supplementation

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Knowledge Level | 2 weeks
  Comparison of mean scores from pre-test and post-test

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Goktas, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No